CLINICAL TRIAL: NCT03752450
Title: Insight in the Development and Recovery of Hypernatremia in Critically Ill Patients.
Brief Title: Prospective Data Analysis of the Development of Hypernatremia in Intensive Care Unit
Acronym: HYPNIC
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Eveline Mestrom, Doctor of Medicine, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: HYPNIC
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Hypernatremia
Keywords: Water-electrolyte imbalance
MeSH Terms: conditions — Hypernatremia; Water-Electrolyte Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: All patients admitted to ICU >48 hours will be included. Eventually, a number of these patients will develop hypernatremia and form the cases. The patients who will not develop hypernatremia will be assigned as the controls.

SUMMARY:
Hypernatremia is frequently encountered in patients admitted to the Intensive Care Unit (ICU) and associated with increased mortality and length of stay. Previous studies focused on predictors in the development and recovery of hypernatremia by including amount and types of administered medication, fluid balance, laboratory results and changes in vital signs. However, data of larger populations or data on infusion rates, fluid and salt balance or renal replacement therapy is lacking. This study aims to provide better insight in the development and recovery of hypernatremia through the collection of detailed information on the input and output of fluids and salts in a larger group of patients than studied before.

DETAILED DESCRIPTION:
Hypernatremia is frequently encountered in patients admitted to the Intensive Care Unit (ICU) and associated with increased mortality and length of stay. The main mechanism is an imbalance between sodium and total body water. Consequently, this poses multiple factors to play a role in the development of hypernatremia. multifactorial. Previous studies focused on predictors in the development of hypernatremia by including amount and types of administered medication, fluid balance, laboratory results and changes in vital signs. However, data of larger populations or data on infusion rates, fluid and salt balance or renal replacement therapy is lacking. Few studies investigated the recovery of hypernatremia, which showed that correction of hypernatremia can reduce the associated mortality risk.

This study aims to provide better insight in the development and recovery of hypernatremia through the collection of detailed information on the input and output of fluids and salts in a larger group of patients than studied before.

ELIGIBILITY:
Inclusion Criteria:

* Adults >17 years old
* Admitted >48 hours in ICU

Exclusion Criteria:

- Expected discharge same day as day of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As a cardiothoracic and oncologic center, the ICU in the Catharina Hospital mostly admits postoperative patients. Other categories of admission are sepsis, respiratory insufficiency, intoxication. However, all patients with an indication for hemodynamic, respiratory of metabolic monitoring will be admitted. The Catharina Hospital is a tertiairy referral hospital. The ICU has 32 beds.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Development of hypernatremia | During ICU admission
  Serum sodium levels >145mmol/L
Recovery of hypernatremia | During ICU admission
  Serum sodium levels returning back to levels below 146mmol/L

SECONDARY OUTCOMES:
Mortality | During ICU admission as well as during hospital admission
  Patient did or did not pass away.
Length of stay | Admission in ICU as well as in hospital
  Number of days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Mestrom, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
If necessary for publication, the data will be provided according to Good Clinical Practice in an anonymized and deidentified fashion.

REFERENCES:
- [Result] Waite MD, Fuhrman SA, Badawi O, Zuckerman IH, Franey CS. Intensive care unit-acquired hypernatremia is an independent predictor of increased mortality and length of stay. J Crit Care. 2013 Aug;28(4):405-12. doi: 10.1016/j.jcrc.2012.11.013. Epub 2013 Jan 29. PMID 23369520
- [Result] Lindner G, Funk GC, Lassnigg A, Mouhieddine M, Ahmad SA, Schwarz C, Hiesmayr M. Intensive care-acquired hypernatremia after major cardiothoracic surgery is associated with increased mortality. Intensive Care Med. 2010 Oct;36(10):1718-1723. doi: 10.1007/s00134-010-1968-4. Epub 2010 Jul 24. PMID 20658124
- [Result] Marshall DC, Salciccioli JD, Goodson RJ, Pimentel MA, Sun KY, Celi LA, Shalhoub J. The association between sodium fluctuations and mortality in surgical patients requiring intensive care. J Crit Care. 2017 Aug;40:63-68. doi: 10.1016/j.jcrc.2017.02.012. Epub 2017 Feb 13. PMID 28347943
- [Result] Bihari S, Festa M, Peake SL, Seppelt IM, Williams P, Wilkins B, Bersten A. Sodium administration in critically ill paediatric patients in Australia and New Zealand: a multicentre point prevalence study. Crit Care Resusc. 2014 Jun;16(2):112-8. PMID 24888281
- [Result] Stelfox HT, Ahmed SB, Zygun D, Khandwala F, Laupland K. Characterization of intensive care unit acquired hyponatremia and hypernatremia following cardiac surgery. Can J Anaesth. 2010 Jul;57(7):650-8. doi: 10.1007/s12630-010-9309-1. Epub 2010 Apr 20. PMID 20405264